CLINICAL TRIAL: NCT04273152
Title: The Potential Role of Advanced Glycation End-products in the Pathogenesis of Paediatric Allergies
Brief Title: Potential Role of AGEs in Paediatric Allergies
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, Professor, Federico II University
Other Study IDs: 176/19
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with allergy: children with allergies
  Interventions: Diagnostic Test: advanced glycation endproducts reader
- healthy control: healthy control (non allergic children)
  Interventions: Diagnostic Test: advanced glycation endproducts reader

INTERVENTIONS:
Diagnostic Test: advanced glycation endproducts reader — advanced glycation endproducts reader

SUMMARY:
Food allergy (FA) is "an adverse health effect arising from a specific immune response that occurs reproducibly" according to the 2010 National Institute of Allergy and Infectious Diseases, National Institutes of Health (NIAID/NIH)-supported Guidelines for the Diagnosis and Management of Food Allergy in the United States (Boyce et al. 2010). Studies have suggested that the natural history of FA has changed during the last two decades, with a dramatic rise in the prevalence, severity of clinical manifestations, and risk of persistence into later ages, leading to an increase in hospital admissions, medical visits, treatments, and burden of care on families and to an important economic impact, with significant direct costs for the families and healthcare system (Skripak et al. 2007; McBride et al. 2012; Gupta et al. 2013). The development of FA might be influenced by genetics, environment, and genome-environment interactions, leading to immune system dysfunction, mediated at least in part by epigenetic mechanisms (Berni Canani et al. 2015; Paparo et al. 2018). Many factors have been postulated to contribute to the onset of FA. Among dietary factors, it has been hypothesized that advanced glycation endproducts (AGEs), present at high level in junk food, could be involved in FA pathogenesis. AGEs are a heterogeneous group of compounds deriving from a non-enzymatic reaction between reducing sugars and free amino groups of proteins, lipids, or nucleic acids. This reaction is also known as the Maillard or browning reaction. The formation of AGEs is a part of normal metabolism, but if excessively high levels of AGEs are reached in tissues and the circulation they can become pathogenic. AGEs are naturally present in uncooked animal-derived foods, and cooking results in the formation of new AGEs within these foods. Consumption of AGE-rich diets is associated with elevated circulating and tissue AGEs and an increase of their pro-inflammatory and pro-oxidant effects. On the other hand, restriction of AGEs prevents inflammation. AGEs not only exert their deleterious actions due to their biological properties, but also through their interaction with specific receptors (RAGE). AGEs are able to activate mast cells and induces a chronic inflammatory state that promotes a Th2 type response. The aim of this study is to evaluate the AGEs levels in FA children compared with healthy controls and subjects with other allergic diseases.

DETAILED DESCRIPTION:
The study is designed to evaluate the AGEs concentration in allergic children compared with healthy controls and to investigate the potential role of AGEs in FA pathogenesis. First, the investigators will define subcutaneous AGEs levels in children affected by allergy, comparing to non-allergy children AGEs levels. Subsequently, the investigators will investigate the possible correlation with dietary habits and the potential effects of AGEs on gut barrier components and on non-immune and immune mechanisms in experimental models.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity
* Both sexes
* Age ≥ 5 and ≤15 years with confirmed diagnosis of allergy (food and/or respiratory), and healthy controls age- and sex-matched.

Exclusion Criteria:

* Non caucasian ethnicity
* Age <5 or >15 years
* Concomitant presence of other chronic diseases not related to allergy (i.e., malignancy, immunodeficiency, cystic fibrosis, celiac disease, autoimmune diseases, neuropsychiatric diseases, diabetes mellitus type 1, chronic inflammatory bowel diseases, malformations of the urinary tract, gastrointestinal tract and/or respiratory tract, genetic-metabolic disorders, nervous system diseases, delayed psychomotor development, chronic lung diseases, hematological diseases)
* Presence of tattoos, scars, moles or lesions on both forearms

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with confirmed diagnosis of allergy and healthy controls consecutively observed at our tertiary center for pediatric allergy will be evaluated for inclusion in the study. Only subjects who will meet the inclusion criteria will be invited to participate in the study. Anamnestic, demographic, anthropometric, and clinical data, as well as information on use of drugs, pre-, pro- or symbiotic products will be collected. Also dietary habits will be evaluated, particularly number, place and time of meals, special diets or elimination diets, frequency of consumption of cereals and derivatives, meat products, fish, eggs, dairy products, fruit and vegetables, legumes, sweets, sweetened beverages and possibly alcoholic drinks and the corresponding cooking methods.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
The advanced glycation endproducts subcutaneous levels | at baseline
  the advanced glycation endproductssubcutaneous levels in allergic children compared with healthy controls.

SECONDARY OUTCOMES:
the correlation between advanced glycation endproducts subcutaneous levels and dietary habits | at baseline
  the correlation between advanced glycation endproducts subcutaneous levels and dietary habits
the investigation of the potential pathogenetic role elicited by AGEs in allergy | at baseline
  * Intestinal permeability (using transepithelial eletrical resistence), tight junction proteins expression (measured as fold change), the epithelial cell-derived danger signal mediators IL-33 and TSLP (pg/ml), RAGE pathway expression (measured as fold change), ROS production (expressed as optical density) analysis on human enterocytes cell line
  * IL-4, IL-5, IL-13, IL-10, IFN-g, IL-6, IL-8, TNF-a determination (pg/ml) on culture supernatants from peripheral blood mononuclear cells
  * Immunohistochemistry analysis of small intestinal biopsies (measured as number of CD25+ mononuclear cells)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Office, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided